CLINICAL TRIAL: NCT00717041
Title: Epidemiology of Depression, Anxiety, and Cognitive Impairment Among Emergency Department Patients
Brief Title: Epidemiology of Depression, Anxiety, and Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Manish Shah, Professor, University of Rochester
Other Study IDs: RSRB 24085; NIH 5K23AG028942
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Depression; Anxiety; Cognitive Impairment
Keywords: Depression; Anxiety; Cognitive Impairment; Emergency medicine; prehospital care
MeSH Terms: conditions — Depression; Anxiety Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Presenting to the ED: Patients who present to the ED

SUMMARY:
Many older adults have undetected health problems and lack basic prevention measures. Failure to identify and treat these conditions can lead to unnecessary morbidity and mortality and a decreased quality of life. Traditional screening and intervention programs, usually based in primary care providers' offices, have been insufficient, particularly in medically underserved populations. Alternate sites for screening and intervention have begun to receive attention and may hold promise.

The emergency department (ED) is the entry point for access to medical and social services for many patients and has the potential to serve as a site to identify older adults with unmet needs. However, we do not know the prevalence of depression and cognitive impairment and how they differ by mode of arrival of the patient to the ED. Second, a question remains as to the validity of screening patients during an acute illness. Upon completion, this study will describe the epidemiology of the population of older adults presenting to the ED.

DETAILED DESCRIPTION:
Many older adults have undetected health problems and lack basic prevention measures. Failure to identify and treat these conditions can lead to unnecessary morbidity and mortality and a decreased quality of life. Traditional screening and intervention programs, usually based in primary care providers' offices, have been insufficient, particularly in medically underserved populations. Alternate sites for screening and intervention have begun to receive attention and may hold promise.

The emergency department (ED) is the entry point for access to medical and social services for many patients and has the potential to serve as a site to identify older adults with unmet needs. However, we do not know the prevalence of depression and cognitive impairment and how they differ by mode of arrival of the patient to the ED. Second, a question remains as to the validity of screening patients during an acute illness. This study aims to:

1. Compare the prevalence of depression and cognitive impairment among patients who arrive at the ED by EMS, as compared to those arriving via other means.
2. Evaluate the reliability of screening patients for depression and cognitive impairment during an acute illness and after the illness.
3. To evaluate correlates of depression, anxiety and suicidal ideation. Upon completion, this study will describe the epidemiology of the population of older adults presenting to the ED.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Arrival at ED

Exclusion Criteria:

* Institutionalized

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All older adults arriving at participating hospital emergency departments to obtain emergency care.
Sampling Method: Non-Probability Sample
Enrollment: 1206 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish N. Shah, MD MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Presenting to the ED
Started | 1206
Completed | 1206
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Presenting to the ED
Number analyzed (Participants) | 1206
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [65 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 634
  Male | 572
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 1184
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 178
  White | 1000
  More than one race | 0
  Unknown or Not Reported | 28
Region of Enrollment [Number; unit: participants]
  United States | 1206
Anxiety (>=10 on GAD7) [Number; unit: participants] — The number of participants with Generalized Anxiety Disorder - 7 scores greater than or equal to 10 (more anxiety).
  participants | 119
Depression (>=10 on PHQ9) [Number; unit: participants] — Number of participants with the Patient Health Questionnaire - 9 (Depression) >= 10 (more depression).
  participants | 177
Cognitive Impairment (>2 on SIS) [Number; unit: participants] — Number of participants with Six Item Screener testing with greater than 2 errors (more errors, worse cognition).
  participants | 106

OUTCOME MEASURES:

1. Primary Outcome: Participants With Depression by Patient Health Questionnaire - 9
Description: Number of participants with depression as measured by the Patient Health Questionnaire - 9, with a score of greater than or equal to 10.
Time Frame: 2 hours
Measure: Number; unit: participants
Arm/Group | Presenting to the ED
Number analyzed (Participants) | 1206
participants | 177

2. Primary Outcome: Participants With Cognitive Impairment by Six Item Screener
Description: Number of participants with cogintiive impairment as measured by the Six Item Screener, with greater than 2 questions incorrect
Time Frame: 2 hours
Measure: Number; unit: participants
Arm/Group | Presenting to the ED
Number analyzed (Participants) | 1206
participants | 106

3. Primary Outcome: Participants With Anxiety by Generalized Anxiety Disorder - 7
Description: Participants with anxiety as measured by the Generalized Anxiety Disorder - 7, with a score greater than or equal to 10.
Time Frame: 2 hours
Measure: Number; unit: participants
Arm/Group | Presenting to the ED
Number analyzed (Participants) | 1206
participants | 119

4. Secondary Outcome: Depression and Cognitive Impairment at 2 Weeks
Description: For the individuals who are able to be contacted in 2 weeks, how many still test positive for depression and cognitive impairment.
Time Frame: 2 weeks
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Depressed in the ED: Patients who present to the ED who test positive for depression
- Cognitively Impaired in the ED: Patients presenting to the ED who have cognitive impairment
Arm/Group | Depressed in the ED | Cognitively Impaired in the ED
Number analyzed (Participants) | 803 | 808
participants | 27 [19 to 38] | 5 [4 to 25]

ADVERSE EVENTS:
Time Frame: While enrolled in the study, 2 weeks
Arm/Group | Presenting to the ED
Serious Adverse Events (participants affected / at risk) | 0/1206
Other Adverse Events (participants affected / at risk) | 0/1206

LIMITATIONS AND CAVEATS:
* Single center, limited generalizability
* Large proportion of individuals lost to follow up
* ED visit may have heightened symptoms
* Validity of instruments in the ED setting is unknown

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No